CLINICAL TRIAL: NCT06433193
Title: Early Feasibility Study to Evaluate the Safety and Efficacy of PAK HD in ESRD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nextkidney S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: DIALYSS-CLI-CIP02
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: End Stage Renal Disease; ESRD
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PAK HD Sorbent Study (Experimental): The study will be performed as a prospective, non-randomised, single arm two-period cross-over study comparing conventional CHD to PAK HD. All adverse events will be recorded and reviewed. Only one subject will enter each study period at a time.
  Interventions: Device: PAK HD Sorbent Therapy

INTERVENTIONS:
Device: PAK HD Sorbent Therapy — Study Period 1:
  Subjects will receive their normal prescribed 4h CHD treatments Monday or Tuesday. On Wednesday or Thursday, one 4h CHD therapy will be performed at a dialysate flow rate (QD) of 300mL/min, identical to the dialysate flow rate of the PAK HD sorbent therapy. Blood and dialysate samples will be collected during treatment and sent for analysis, for comparison with PAK HD sorbent treatment.
  Study Period 2:
  Subjects will again receive their normal prescribed 4h CHD treatments Monday or Tuesday. On Wednesday or Thursday, a 2h PAK HD +/- 2h CHD therapy will be performed. Blood and dialysate samples will again be collected during treatment and sent for analysis, for comparison with the CHD therapy of the first period. After completion of study period 2 (PAK HD +/- CHD), subjects will be observed for a minimum duration of 1 h in the hospital after which they may go home if the post-dialysis period was uneventful.

SUMMARY:
The purpose of this study is to demonstrate the safety of dialysate regeneration of the PAK HD sorbent cartridge and therapy efficacy of the PAK HD sorbent therapy compared with conventional hemodialysis.

DETAILED DESCRIPTION:
This clinical trial is being conducted to evaluate the biochemical safety of dialysate regeneration with the PAK HD sorbent cartridge in a limited number of patients and treatments. Therapy efficacy of the PAK HD sorbent therapy will be compared to conventional hemodialysis under the same therapy settings. The trial will use only one single PAK HD sorbent therapy per patient, and a total of 3 patients. The PAK HD therapies will be performed in the middle of the week.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be adults >/= 21 years old and <80 years old.
2. Subjects must be weighing >/= 55kg and <90kg (patient's dry weight).
3. Subjects must have stable haemoglobin >/= 10.5g/dL, 2 months prior to enrolment
4. Subjects' pre-dialysis serum values must be within the following range, 2 months prior to enrolment:

   Patient allowable serum biochemistry ranges Allowable pre-dialysis serum values Na >/= 132 mmol/L or </= 145mmol/L HCO3 >/= 15mmol/L or </= 30mmol/L K >/= 3.5mmol/L or </= 5.8mmol/L
5. Subjects on stable on thrice weekly 4-h HD schedule. Stability is defined as:

   * Haemodynamic stability during dialysis (absence of hypotensive events and symptomatic arrhythmias), no angina pectoris, AND
   * No altered level of consciousness during dialysis.
6. Subjects with a well-functioning vascular access (native fistula graft):

   * capable of providing a blood flow rate of >/= 250 mL/min, AND
   * no vascular access revision and stable shunt flow for at least 4 weeks prior to enrolment.
7. Subjects capable of understanding the informed consent form and give informed consent.
8. Subjects willing and able to comply with study procedures and to attend all study follow-up visits.
9. Subjects who are female of reproducible age to practice birth control methods.
10. Subjects can be either gender.

Exclusion Criteria:

1. Subjects with haemoglobin level of <10.5g/dL in any measurement 2 months prior to enrolment.
2. Subjects with the following pre-dialysis serum values in any measurement 2 months prior to enrolment:

   * sodium concentration <132 mmol/L or > 145mmol/L
   * bicarbonate <15mmol/L or >30mmol/L
   * plasma potassium concentration <3.5mmol/L or >5.8mmol/L
   * urea <15mmol/L or >28 mmol/L
3. Subjects with severe hypertension: systolic blood pressure > /=180 mmHg, diastolic blood pressure >/=120 mmHg in any officemeasurement less than 4 weeks prior to enrolment.
4. Subjects with chronic obstructive pulmonary disease or any respiratory disease that may predispose to CO2 retention.
5. Subjects with impaired liver function. Impaired liver function is defined as an elevated ALT (alanine aminotransferase) by 3-fold orgreater above the upper limit of normal.
6. Subjects with episodes of haemolysis in any measurement 3 months prior to enrolment.
7. Subjects with a central venous catheter.
8. Subjects with vascular access dysfunction (whether or not requiring an intervention), i.e. failure to achieve and/ or sustain a bloodflow of >/=250 mL/min and/or signs of compromised vascular access patency (according to the opinion of the investigator) within 4weeks prior to enrolment.
9. Subjects with vascular access related infection less than 4 weeks prior to enrolment
10. Subjects requiring an average ultrafiltration volume >2.8 L per 4-h treatment in mid-week dialysis session in the past 4 weeks priorto enrolment.
11. Subjects who are on heparin free dialysis
12. Subjects who are unable to provide informed consent.
13. Subjects who are unable to comply with study procedures.
14. Subjects with psychosocial problems which may negatively influence dialysis treatment.
15. Subjects who participated in another clinical intervention or device trial less than 12 weeks prior to enrolment, are currentlyparticipating or intend to participate in such a trial.
16. Subjects who are pregnant, breast feeding, or planning a pregnancy within the study period.
17. Subjects with a life expectancy <1 year.
18. Subjects who are anticipating a living donor kidney transplantation within < 2 months of the study period.
19. Subjects with recent history of drug and/or alcohol abuse in the last 3 months prior to enrolment.

Ages: 21 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2024-02-22 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
The primary objective of this early feasibility clinical trial is to assess the (short term) clinical safety of the PAK HD sorbent treatment in a limited number of patients and treatments. | 2 weeks
  The clinical safety of the PAK HD will be evaluated in terms of the following primary endpoints:
  1. Absence of serious adverse events (SAE)
  2. Absence of critical change in patient's clinical condition and vital parameters (Blood pressure, heart rate, body temperature and respiratory rate and pulse oximetry) during treatment.
  3. Absence of critical change in haematology and biochemistry immediately before the start of therapy and immediately after completion of therapy, including acid-base state, electrolytes, and ammonia.

SECONDARY OUTCOMES:
The secondary objective of this study is to evaluate the efficacy of the PAK HD therapy in comparison to CHD, in terms of uremic toxin removal efficacy (urea, creatinine and phosphate). | 2 weeks
  The therapy efficacy will be evaluated with the secondary endpoint:
  a) PAK HD therapy provides equivalent toxin clearances for urea, phosphate and creatinine as compared to CHD

CONTACTS AND LOCATIONS:
Overall Officials: Titus Wai Leong Lau, MD, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital Investigational Medicine Unit, Singapore, Singapore